CLINICAL TRIAL: NCT03031587
Title: Validation of Thermometric Cardiac Imaging by MRI
Acronym: VAIMTH-IRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2016/15
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2020-02

CONDITIONS: Cardiac MRI
Keywords: Thermometric MRI; Myocardium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI examination (Experimental): Each patient coming to the hospital for cardiac MRI examination can participate to the study if he/she meets the eligibility criteria
  Interventions: Other: Additional MRI acquisition sequences; Device: MRI

INTERVENTIONS:
Other: Additional MRI acquisition sequences — It deals with specific sequences of rapid imaging acquisition in gradient echo (4 to 5 slices/cardiac cycle) with synchronization on the surface ECG systematically included in a cardiac MRI examination, together with update of the slice position depending on the respiratory state (established technique of navigator echo). The acquisition is repeated over 300 cardiac cycles to monitor myocardial temperature changes
Device: MRI — cardiac MRI

SUMMARY:
Radiofrequency ablation is the primary treatment for atrial and ventricular arrhythmias resistant to medication. However, the absence of assessment of injury creation during radiofrequency application is an important issue. One of the objectives of the Institut Hospitalo-Universitaire (IHU) Liryc (l'Institut de Rythmologie et Modélisation Cardiaque) is to improve ablation procedures by radiofrequency of cardiac arrhythmias. This is based on thermometric imaging by Magnetic Resonance Imaging (MRI) which allows a real time visualization of tissue temperature in all the myocardium with sufficient spatial and temporal resolution to characterize the induced thermal lesion. Today, investigators have developed and validated a new method for cardiac thermometry, associating rapid MRI acquisition technique (4 to 5 slices per heart beat) with online image reconstruction and correction algorithms against residual motion, magnetic susceptibility, drift of the magnetic field, etc... Recent preclinical studies showed a precision of 1°Celsius in the myocardium, largely sufficient to characterize a thermal treatment induced by radiofrequency where typical temperature rises of 40°C are observed during ablation. Temporal evolution of the temperature in each pixel provides access to calculation of the accumulated thermal dose that is a relevant indicator of the induced necrosis.

This imaging method must now be evaluated in humans in order to test its robustness under real conditions (presence of arrhythmias, corpulent patients, etc…) and to optimize acquisition parameters and image processing. The aim of this research is thus to obtain specific MRI sequence of images of patients, on which will be evaluated the different algorithms of reconstruction and processing for temperature imaging. This study is a mandatory step in the perspective of future clinical treatments of cardiac arrhythmia under MRI.

DETAILED DESCRIPTION:
Radiofrequency ablation is the primary treatment for atrial and ventricular arrhythmias resistant to medication. However, the absence of assessment of injury creation during radiofrequency application is an important issue in that it can result either in recurrences of arrhythmia requiring redo procedures when an inadequate lesion is created, or on the opposite in serious complications when the lesion created is too large and extents to extra-cardiac territory that should be preserved. The imaging team of the IHU-Liryc develops new methods in cardiac MRI in view of diagnostics (improve spatial and temporal resolution, dynamic 3D imaging or contrast improvement) and therapeutics. Hence, one of the objectives of the IHU-Liryc is to improve ablation procedures by radiofrequency of cardiac arrhythmias in order to make them more effective (Real-time visualization of the thermal lesion, allowing application of the sufficient energy needed for a transmural lesion), and safer avoiding excessive lesion responsible for perforation and extension to extra-cardiac structures. This is based on thermometric imaging by MRI which allows a real time visualization of tissue temperature in all the myocardium with sufficient spatial and temporal resolution to characterize the induced thermal lesion. MRI thermometry was developed during the last decade and successfully applied clinically over a wide range of organs (the uterus, the brain, the liver, the kidneys) for direct monitoring of thermal treatment of various pathologies (fibroids Uterus, bone metastasis, liver cancer). This innovative technic was not applicable to cardiac arrhythmias due to the respiratory and cardiac movements whose rhythms can be irregular, as well as thermal noise generated by blood flow on images. Today, our team has developed and preclinically validated a new rapid MRI method dedicated to cardiac thermometry. All patients who give their oral agreement to participate to the study will have added to their examination some acquisition sequences. The maximum additional time due to the specific acquisitions of the study will be 5 minutes, over an average clinical examination time of 45 minutes. No follow-up or visit of end of treatment will be performed, the end of patient participation in this research corresponding to the end of the MRI examination.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring, as part of his/her traditional management of an MRI imaging examination
* Adults (age greater than or equal to 18 years) of both sexes
* Minors (aged 15 to 18) of both sexes subject to the parental agreement or its legal representative
* Patient's oral agreement after reading the information note
* Patient affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* Patients under 15 years of age
* Patient unable to give oral consent
* Patients in periods of relative exclusion in relation to another protocol
* Patient deprived of liberty by judicial or administrative decision
* Major protected by the law
* Patient who does not meet the eligibility criteria for an MRI examination with or without injection.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Calculation of the temperature variance of various measurements realized in a region of interest of the myocardium | Day 0
  1 measurement of temperature (°C) by cardiac beating

CONTACTS AND LOCATIONS:
Overall Officials: Pierre JAÏS, MD PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No